CLINICAL TRIAL: NCT07380256
Title: Effects of Impaired Visual Acuity and Binocular Control Abnormalities (VABC) on Vestibulo-ocular Reflex (VOR) Adaptation in Adults With and Without Vestibular Hypofunction
Brief Title: Visual Influences on Vestibular Adaptation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Colin R. Grove, Assistant Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2025P012555
Record Dates: First submitted 2026-01-20; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Vestibular Hypofunction; Binocular Vision Abnormalities; Reduced Vision
Keywords: vestibulo-ocular reflex; incremental vestibulo-ocular reflex adaptation; abnormal uncorrected static visual acuity; Gait Disorientation Test; video head impulse test; vertical and torsional alignment nulling; dynamic visual acuity test; modified Clinical Test of Sensory Interaction in Balance
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Intervention Model Description: This study uses a prospective, cross-over observational design in which participants complete two sessions of incremental vestibulo-ocular reflex adaptation (IVA) under different visual conditions. Participants are assigned to one of four groups based on visual status and vestibular function (abnormal visual acuity, binocular vision abnormalities, with or without vestibular hypofunction).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: Abnormal Uncorrected Static Visual Acuity (No Vestibular Hypofunction) (Experimental): Adults with abnormal uncorrected distance visual acuity and normal vestibular function.
  This group will be part of Experiment 1. This experiment studies people whose main visual problem is reduced uncorrected distance visual acuity (i.e., blurry vision without glasses/contacts).
  Experiment 1 tests the effect of blurry vision on VOR adaptation
  Interventions: Other: Incremental Vestibulo-Ocular Reflex Adaptation (IVA)
- Group 2: Abnormal Uncorrected Static Visual Acuity + Vestibular Hypofunction (Experimental): Adults with abnormal uncorrected distance visual acuity and unilateral vestibular hypofunction.
  This group will be part of Experiment 1. This experiment studies people whose main visual problem is reduced uncorrected distance visual acuity (i.e., blurry vision without glasses/contacts).
  Experiment 1 tests the effect of blurry vision on VOR adaptation
  Interventions: Other: Incremental Vestibulo-Ocular Reflex Adaptation (IVA)
- Group 3: Binocular Vision Abnormalities (No Vestibular Hypofunction) (Experimental): Adults with binocular vision abnormalities (e.g., convergence insufficiency, ocular misalignment) and normal vestibular function.
  This group will be part of Experiment 2. This experiment studies people whose main visual problem is how the two eyes work together (e.g., convergence insufficiency, ocular misalignment).
  Experiment 2 tests the effect of binocular vision dysfunction on VOR adaptation
  Interventions: Other: Incremental Vestibulo-Ocular Reflex Adaptation (IVA)
- Group 4: Binocular Vision Abnormalities + Vestibular Hypofunction (Experimental): Adults with binocular vision abnormalities and unilateral vestibular hypofunction.
  This group will be part of Experiment 2. This experiment studies people whose main visual problem is how the two eyes work together (e.g., convergence insufficiency, ocular misalignment).
  Experiment 2 tests the effect of binocular vision dysfunction on VOR adaptation
  Interventions: Other: Incremental Vestibulo-Ocular Reflex Adaptation (IVA)

INTERVENTIONS:
Other: Incremental Vestibulo-Ocular Reflex Adaptation (IVA) — IVA is delivered using the StableEyes device, which includes a lightweight head-mounted unit with inertial sensors and a micromirror that controls the position of a low-power laser target projected onto a wall. The device adjusts the target's movement based on the participant's head velocity to create a controlled visual error signal that induces vestibulo-ocular reflex (VOR) adaptation. During each session, participants sit about one meter from a blank wall and perform rapid, self-generated head impulses while visually tracking the moving laser target. The target appears at neutral, moves at a fraction of head velocity during each impulse, and briefly disappears before reappearing at center. Each session lasts 15 minutes and includes roughly 150 head impulses in the horizontal or vertical plane. The procedure has been well-tolerated in prior studies with no reported adverse events.

SUMMARY:
The goal of this study is to determine whether impaired static visual acuity or binocular vision abnormalities affect vestibulo-ocular reflex (VOR) adaptation in adults with and without vestibular hypofunction.

The main questions it aims to answer are:

* Does reduced static visual acuity change the amount of VOR adaptation achieved during incremental VOR adaptation (IVA) training?
* Do binocular vision abnormalities limit VOR adaptation in otherwise healthy adults or in adults with vestibular hypofunction?

Because this study includes comparison groups, researchers will compare participants with normal vestibular function and impaired visual acuity versus those with abnormal vestibular function and impaired visual acuity, as well as participants with normal vestibular function and binocular vision abnormalities versus those with abnormal vestibular function and binocular vision abnormalities, to determine whether these visual conditions affect the magnitude of VOR gain change following IVA training.

DETAILED DESCRIPTION:
Impairment of vestibular pathways can lead to deficits in balance, gait, and gaze stability. Gaze-stability exercises are a central component of vestibular rehabilitation and have been shown to improve vision during head movement as well as functional mobility in individuals with peripheral or central vestibular dysfunction. Improvements in gaze stability may occur through vestibulo-ocular reflex (VOR) adaptation or through compensatory saccadic eye movements. However, many adults with vestibular hypofunction also present with uncorrected visual acuity deficits or binocular vision abnormalities, such as low vision, convergence insufficiency, or ocular misalignment. These visual conditions are common but understudied in the context of vestibular rehabilitation, and it is not known whether they limit the capacity for VOR adaptation.

Incremental vestibulo-ocular reflex adaptation (IVA) is a non-invasive, 15-minute training method that strengthens the VOR by exposing users to a controlled visual error signal. IVA uses a moving laser target whose velocity is programmed as a function of the participant's head movement, producing immediate increases in VOR gain. The method can be customized to provide unilateral, bilateral, or asymmetric adaptation, allowing targeted training for individuals with unilateral or bilateral vestibular deficits. IVA has been studied extensively in adults with vestibular hypofunction, but its effectiveness in individuals with impaired visual acuity or binocular vision abnormalities has not been evaluated.

This study will examine whether reduced static visual acuity or binocular vision abnormalities affect the magnitude of VOR adaptation in adults with and without vestibular hypofunction. Two experiments will be conducted using a cross-over design. Experiment 1 will enroll adults with abnormal uncorrected static visual acuity, with and withoutvestibular hypofunction, to compare VOR adaptation with and without vision correction. Experiment 2 will enroll adults with binocular vision abnormalities, with and without vestibular hypofunction, to evaluate VOR adaptation in their best corrected visual state. All participants will complete IVA training during two study visits separated by a washout period.

ELIGIBILITY:
Inclusion Criteria:

For All Participants (All Groups)

* Age 18 to 89 years
* Able to provide informed consent

Group-Specific Inclusion Criteria Group 1: Abnormal Uncorrected Static Visual Acuity (No Vestibular Hypofunction)

* Abnormal uncorrected distance visual acuity based on LogMAR thresholds
* No clinical evidence of vestibular hypofunction on vHIT

Group 2: Abnormal Uncorrected Static Visual Acuity + Vestibular Hypofunction

* Abnormal uncorrected distance visual acuity
* Vestibular hypofunction confirmed by vHIT (reduced lateral canal gain and corrective saccades)

Group 3: Binocular Vision Abnormalities (No Vestibular Hypofunction)

* Presence of binocular vision abnormalities (e.g., convergence insufficiency, ocular misalignment)
* No vestibular hypofunction on vHIT

Group 4: Binocular Vision Abnormalities + Vestibular Hypofunction

* Binocular vision abnormalities as above
* Vestibular hypofunction confirmed by vHIT

Exclusion Criteria:

* Neurological disorders affecting eye movements or balance (e.g., stroke, multiple sclerosis, Parkinson's disease)
* History of traumatic brain injury
* Active or unstable medical conditions that could interfere with participation
* Uncorrected hearing impairment that prevents following instructions
* Inability to perform repeated head impulses due to cervical spine, musculoskeletal, or pain limitations
* Current use of medications that significantly affect vestibular function (e.g., vestibular suppressants)
* Prior vestibular surgery
* Severe visual impairment not correctable with lenses
* Pregnancy (due to balance testing requirements)
* Any condition that, in the investigator's judgment, would interfere with safe participation

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in Vestibulo-Ocular Reflex (VOR) Gain | Baseline (visit 1) (before and after after IVA intervention), Visit 2 (2-10 days from baseline) (before and after IVA intervention)
  VOR gain will be measured using the video head impulse test (vHIT). Gain is calculated as eye velocity divided by head velocity during high-acceleration, moderate velocity, small amplitude head rotations in the plane of the semicircular canals. This outcome quantifies the strength of the vestibulo-ocular reflex, with higher gain values indicating stronger VOR responses, with normal gain = 0.8 to 1.2. The change in VOR gain from before to after training will be used to assess VOR adaptation.
  IVA: Incremental Vestibulo-Ocular Reflex Adaptation

SECONDARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | Baseline (Visit 1)(pre IVA intervention), Visit 2 (2-10 days from baseline)(pre IVA intervention)
  A 25-item questionnaire assessing perceived handicap due to dizziness. Total score ranges from 0 to 100, with higher scores indicating greater perceived disability.
Visual Vertigo Analogue Scale (VVAS) | Baseline (Visit 1)(pre IVA intervention), Visit 2 (2-10 days from baseline)(pre IVA intervention)
  Nine visual-vertigo provoking scenarios rated on a 0-10 scale. A total score is calculated by averaging completed items and multiplying by 10. Higher scores indicate more severe visually induced dizziness.
Oscillopsia Visual Analog Scale (OVAS) | Baseline (Visit 1)(pre IVA intervention), Visit 2 (2-10 days from baseline) (pre IVA intervention)
  Participants rate the severity of unstable vision during head movement while walking 20 feet. Scores are transformed to a 0-100 scale, with higher scores indicating more severe oscillopsia.
Disequilibrium Visual Analog Scale (DVAS) | Baseline (Visit 1)(pre IVA intervention), Visit 2 (2-10 days from baseline)(pre IVA intervention)
  Participants rate the severity of imbalance while walking 20 feet. Scores are transformed to a 0-100 scale, with higher scores indicating greater disequilibrium.
Change in Modified Clinical Test of Sensory Interaction in Balance (mCTSIB) | Baseline (visit 1) (before and after after IVA intervention), Visit 2 (2-10 days from baseline) (before and after IVA intervention)
  Participants stand under four sensory conditions (eyes open/closed on firm/foam surfaces). Outcomes include time maintained (0-120 seconds) and postural sway metrics from inertial measurement units. Higher times indicate better balance.
Change in Gait Disorientation Test (GDT) | Baseline (visit 1) (before and after after IVA intervention), Visit 2 (2-10 days from baseline) (before and after IVA intervention)
  Participants walk 20 feet with eyes open and eyes closed. The GDT score is the difference in time between the two conditions. Larger differences indicate greater gait disorientation.
Dynamic Visual Acuity Test (DVAT) | Baseline (Visit 1)(pre IVA intervention), Visit 2 (2-10 days from baseline)(pre IVA intervention)
  Difference between static visual acuity and best dynamic visual acuity (LogMAR) during active head impulses to the right and left. Larger differences indicate poorer dynamic visual acuity.
Vertical Alignment Nulling (VAN) and Torsional Alignment Nulling (TAN) | Baseline (Visit 1)(pre IVA intervention), Visit 2 (2-10 days from baseline)(pre IVA intervention)
  Participants align dichoptic red and blue lines in a virtual environment. The absolute deviation from true alignment provides a measure of vertical or torsional ocular misalignment. Larger deviations indicate greater misalignment.
Compensatory Saccade Metrics | Baseline (Visit 1)(pre IVA intervention), Visit 2 (2-10 days from baseline) (pre IVA intervention)
  Frequency, latency, amplitude, and accuracy of covert and overt compensatory saccades during vHIT. These metrics characterize compensatory eye-movement strategies associated with vestibular hypofunction.
Activities-specific Balance Confidence Scale (ABCS) | Baseline (Visit 1)(pre IVA intervention), Visit 2 (2-10 days from baseline)(pre IVA intervention)
  A 16-item self-report measure of balance confidence in daily activities. Scores range from 0% (no confidence) to 100% (complete confidence). Higher scores indicate greater balance confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Grove, PT, DPT, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Ophthalmology Clinics, Atlanta, Georgia
  - Dizziness and Balance Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
A complete de-identified dataset will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after the primary outcome is published; indefinitely
Access Criteria: Mechanism: Through the Open Science Framework or Emroy Dataverse